CLINICAL TRIAL: NCT00845286
Title: Investigation of Myocardial Function and Vascular Adaptation in Association With Genotype in Marathon Runners
Brief Title: Marathon, Genetics, Inflammation and the Cardiovascular System: MAGIC-Trial
Acronym: MAGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1807/07-II
Record Dates: First submitted 2008-09-19; First posted 2009-02-18 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure; Sudden Cardiac Death
Keywords: exercise, myocardial dysfunction, endothelial dysfunction,; polymorphism
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac; Motor Activity | interventions — Magic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Munich Marathon — 42,195 km marathon run
  Other Names: MAGIC

SUMMARY:
The purpose of the study is to determine the myocardial function and vascular adaptation after strenuous exercise in association with genotype/polymorphisms. We aim to investigate the effects of extreme endurance exercise on the cardiovascular system. Furthermore, the role of the inflammatory response and adaptive mechanisms of the vasculature are examined. Subclinical injuries to the myocardium and vascular wall are being investigated.

DETAILED DESCRIPTION:
Regular exercise leads to an improvement of cardiovascular risc factors in patients with coronary heart disease, atherosclerosis and metabolic disorders. Aerobic exercise has anti-inflammatory effects. In contrast, the exertional exercise of marathon running causes an acute pro-inflammatory impulse. This may lead to myocardial injury and, in case of preexisting plaques, may result in plaque rupture and acute myocardial infarction.

We aim to define the critical role of inflammatory markers and cardiovascular risc factors as a predictor of an increased risk for myocardial and endothelial dysfunction in marathon runners.

Diagnostic tools include measurements of augmentation index (AIx), arteriolar-venular ratio (AVR) and, for the first time, 2D and 3D echocardiographic measurements such as TDI-imaging and speckle tracking. Inflammatory markers include c-reactive protein (CRP), interleukins and tumor necrosis factor. Additionally, cardiovascular markers are measured. All variations are analysed on the basis of genotype characteristics/polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* men aged 30-60 years

Exclusion Criteria:

* manifested heart disease
* insulin dependent diabetes mellitus
* multi drug therapy
* GFR<60ml/min.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2008-09; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
E/A ratio | pre-, post-, one day follow-up

SECONDARY OUTCOMES:
LV twist | pre-, post-, one day follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prevention and Sports medicine, Munich, Bavaria, Germany